CLINICAL TRIAL: NCT07335848
Title: The Effect of Physical Activity Cards Adapted With Life Kinetik Exercises on Cognitive Functions and Problem-solving Skills in Middle School Students: a Randomized Controlled Trial
Brief Title: Cognitive Effects of Life Kinetik-Adapted Physical Activity Cards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enes Sucular (Other)
Responsible Party: Sponsor-Investigator, Enes Sucular, Principal Investigator, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 230037-77
Record Dates: First submitted 2025-12-30; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Childeren; Life Kinetik; Students; Physicial Activity; Excercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Life Kinetik Group (Experimental): Participants in this group took part in an intervention involving physical activity cards adapted with Life Kinetik exercises three times a week for 12 weeks. The training program combined physical and cognitive tasks designed to improve cognitive functions and problem-solving skills.
  Interventions: Behavioral: Life Kinetik Adapted Physical Activity Cards Training
- Fiziksel Activity Group (Experimental): Participants in this group took part in an intervention involving physical activity cards three times a week for 12 weeks. The training program combined physical and cognitive tasks designed to assess its effect on cognitive functions and problem-solving skills.
  Interventions: Behavioral: Physical activity cards training
- Control Group (No Intervention): Participants in the control group continued their normal daily lives without any additional intervention. To provide an environment equivalent to the experimental group's exposure, they participated in structured games unrelated to the goals of Life Kinetik and Physical Activity Cards. These activities included light stretching movements and educational games. They were conducted at the same frequency and duration as the experimental sessions (three times a week for one hour). At the end of the study, participants were fully informed about the nature and purpose of their activities, including the rationale for the placebo-like design, as part of the ethical protocol.

INTERVENTIONS:
Behavioral: Life Kinetik Adapted Physical Activity Cards Training — A combination of cognitive and physical exercises aimed at developing cognitive functions and problem-solving skills.
  Arms: Life Kinetik Group
Behavioral: Physical activity cards training — Cards used in physical education classes in Turkish middle schools that include movement skills aimed at improving physical fitness.
  Arms: Fiziksel Activity Group

SUMMARY:
The purpose of this study is to investigate the effects of physical activity cards integrated with Life Kinetik exercises on attention, short-term memory, cognitive flexibility, and problem-solving skills in middle school students. The study specifically aims to determine whether this integrated educational approach leads to greater improvements in cognitive performance compared to traditional physical activity cards.

DETAILED DESCRIPTION:
This study evaluated the effects of physical activity cards adapted with Life Kinetik exercises on cognitive functions and problem-solving skills in middle school students. A total of 36 participants aged 11-14 years were assigned to two experimental groups (physical activity cards adapted with Life Kinetik and physical activity card) and one control group in a 12-week intervention designed with a pre-test-post-test experimental model. The PAC-LK group participated in physical activity cards integrated with Life Kinetik exercises, while the physical activity card group followed traditional physical activity cards, each conducted three times per week for one hour, and the control group did not receive any intervention. The integrated program combined physical movement with cognitive tasks to stimulate cognitive processing and executive functions. Outcome measures included attention, short-term memory, cognitive flexibility, and problem-solving performance.

ELIGIBILITY:
Inclusion Criteria:

* Secondary school pupils aged 11 to 14,be enrolled in secondary school,Healthy participants with no chronic illnesses, musculoskeletal injuries, or physical limitations in the last six months.

Exclusion Criteria:

* To be included in an individualised education programme (IEP), Loss of senses such as hearing or sight, Insufficient Turkish reading comprehension skills.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Stroop test TBAG form | 12 week
  The Stroop Test TBAG Form, physical activity cards adapted with Life Kinetik and physical activity card intervention programmes were used to evaluate their effects on attention and executive functions. The test was specifically applied to assess executive function components that measure focused and selective attention, resistance to distracting stimuli, and information processing speed. The test includes sections such as the Stroop interference score, test speed factor, total time, total number of errors, and total number of corrections. These sections were evaluated to examine the effect on attention and cognitive control processes.The completion time for each section of the test is recorded in seconds. As the time decreases, the performance shown on the test increases. The Stroop Test TBAG Form was developed as part of the BILNOT Battery, a measurement tool with proven validity and reliability, supported by the TÜBİTAK Basic Sciences Research Group.
Visual Auditory Number Sequences Test Form B | 12 week
  The Visual-Auditory Number Sequences Test Form B (VANST-B) was used to assess short-term attention and memory capacity. The test was administered to examine the impact of the physical activity cards adapted with Life Kinetik and physical activity card intervention programs on short-term attention and memory performance. The test includes auditory stimulation, visual stimulation, verbal expression, written explanation, and test total score sections. These sections were evaluated to examine their effects on short-term attention and memory. Before the test, the participants were informed about the application procedure and given a brief trial. Scoring was based on the longest sequence that the participant could correctly repeat.The lowest score obtained in the test is 0, and the highest score is 36. As the score increases, performance improves. The VANST-B is a valid and reliable measurement tool used to assess attention and memory capacity in children.
Cognitive Flexibility Scale | 12 week
  The Cognitive Flexibility Scale (CFS) was used to assess participants' levels of cognitive flexibility. Total scores obtained from the scale were analyzed to determine the effect of the physical activity cards adapted with Life Kinetik and physical activity card intervention programs on cognitive flexibility. This measurement tool is a 6-item Likert-type scale consisting of 12 items and a single subscale. High scores indicate that individuals have high levels of cognitive flexibility, while low scores indicate that they have low levels of cognitive flexibility.
Problem solving inventory for elementary school children | 12 week
  The Problem Solving Inventory for Children at the Primary School Level was used to assess children's problem-solving skills. The total scores obtained from the inventory were analyzed to examine the effects of physical activity cards adapted with Life Kinetik and physical activity card interventions on problem-solving skills.This measurement tool is a 5-point Likert-type scale consisting of 24 items and a single sub-dimension. High scores indicate that individuals have high problem-solving skills, while low scores indicate that problem-solving skills are low.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University Faculty of Sports Sciences, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to ensure the privacy and confidentiality of participants. Additionally, explicit consent for data sharing was not obtained from participants or their guardians during the study, and the ethical approval did not include provisions for sharing individual data externally.